CLINICAL TRIAL: NCT06398847
Title: An Open-label Study of Self-hypnosis Software for Virtual Reality for the Treatment of HIV-associated Chronic Pain - a Development and Usability Study
Brief Title: Virtual Reality (VR) Self-Hypnosis Software
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mary Catherine George, Director Clinical Research, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY-23-00989; GCO#21-1216 (Other Grant/Funding Number: i Prism Grant)
Record Dates: First submitted 2024-03-28; First posted 2024-05-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Musculoskeletal Pain; Neuropathic Pain; Neuralgia
Keywords: HIV chronic pain; Self-hypnosis; virtual reality software; non-drug treatment for chronic pain
MeSH Terms: conditions — Musculoskeletal Pain; Neuralgia

STUDY DESIGN:
Intervention Model Description: This is a combination device of virtual software developed by the study team to be inserted into an off the shelf virtual reality headset.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HIV-associated Chronic Pain Patients (Other): The participants will be enrolled into an open label arm to determine feasibility and useability of the combination device.
  Interventions: Device: Virtual Reality headset

INTERVENTIONS:
Device: Virtual Reality headset — Self-hypnosis software in a Virtual Reality headset. This is the development of software that provides a self-hypnosis experience that can be inserted into any virtual reality device.
  Other Names: OculusGo™

SUMMARY:
This single-site study of self-hypnosis software using an off-the-shelf virtual reality (VR) device (OculusGo™) to determine the software's safety, usability, and preliminary efficacy in pain relief for HIV-associated chronic pain patients. This is funded under the i Prism Funding through Mount Sinai Innovations.

DETAILED DESCRIPTION:
The study will be done in two phases - Phase A is the development of the software by the study team and the engineers targeted to be completed by 4/15/2024. Testing will occur with only the study team. No participants will be involved in the testing phase. Phase B is the participant enrollment phase targeted to start 5/20/2024. A request for FDA Exemption of a non-significant risk combination device has been submitted and granted.

ELIGIBILITY:
Patient Eligibility

Inclusion Criteria:

* Adults age ≥18
* Confirmed diagnosis of HIV, currently on a stable antiretroviral regimen ≥ 90 days.
* Documentation of chronic pain associated with HIV for≥90 days
* Stable pain management regimen ≥90 days, or no pain treatments ≥90 days
* Average pain intensity of 3 or greater on the NRS of the mean daily scores reported between Visit 1 and Visit 2
* Access to the internet via smartphone, computer, or tablet 7. Fluent in English
* Capable of giving informed consent and willingness to comply with study procedures.

Exclusion Criteria:

* A co-occurring medical or psychiatric condition which would make participation in the study or complicate measurement of changes associated with the intervention.
* Concurrent participation in another investigational protocol for pain treatment
* A psychiatric disorder, medical condition, or other life circumstance, which in the opinion of the PI, would contraindicate attendance at sessions, or make it unlikely that the participant could successfully complete the study procedures.
* Current or prior diagnosis of epilepsy, seizure disorder, dementia, migraines, or other neurological conditions contraindicating the use of virtual reality devices.
* A medical condition predisposing prospective participant to nausea or dizziness 6. Lack of stereoscopic vision or severe hearing impairment
* Injury to eyes, face, or neck that impedes using the VR device
* If participant has access to personal VR gear for gaming or other purposes at home, participant fails to agree not to use these personal VR gear during the course of the protocol.
* Currently pregnant or planning to become pregnant during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of times the software is used | twenty one days
  Feasibility of self-hypnosis software using VR devices as measured by frequency of use. The device software will have an ability to determine the number of times each participant used the self-hypnosis software during the 21-day period.
Number of adverse events related to the device | twenty one days
  Safety will be measured by any adverse events related to the use of the software and the device.

SECONDARY OUTCOMES:
Quality of Life measured using Pain, Enjoyment and General Activity Scale (PEG) | at Week 2, 3 and week 4
  Participants perception of pain and quality of life will be measured using the Pain, Enjoyment and General Activity Scale (PEG). The PEG (pain, enjoyment, general activity) composite score will be used to assess pain intensity and interference. The PEG is a 3-item score with potential responses of 0 to 10 with 10 being the most severe pain. The 3 PEG items referring to the past week are: average pain, how pain interfered with enjoyment of life, how pain interfered with general activity To compute the PEG score, add the responses to the questions above, then divide by three to get a final score out of 10, full scale ranges 0 (no pain) to 10 (most severe pain), with higher scores indicate higher levels of pain.
Quality of life measured using Short Form Brief Pain Inventory (SF-BPI) Scale | at Week 2, 3 and week 4
  Participants perception of pain and quality of life will be measured using the Short Form Brief Pain Inventory (SF-BPI) Scale. BPI-SF is a 9-item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. This is a 10-point scale with 0 being the best possible score, meaning "no pain", and 10 being the worst possible score, meaning "pain as bad as you can imagine", thus, higher scores indicate worse health outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: CSR
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  To achieve aims in the approved proposal. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in the University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link to be determined).